CLINICAL TRIAL: NCT02907268
Title: A Single Blind, Split-Face, Randomized, Pilot Study Comparing the Effects of Intradermal and Intramuscular Injection of Two Commercially Available Botulinum Toxin A Formulas to Reduce Signs of Facial Aging
Brief Title: Botulinum Toxin A Single Blind Split-Face Randomized Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ICLS Dermatology & Plastic Surgery (Other)
Responsible Party: Principal Investigator, Sheetal Sapra, Director of Dermatology, ICLS Dermatology & Plastic Surgery
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ICLS-06-2013
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Facial Rhytids
Keywords: botulinum toxin type A, intradermal
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm A (Active Comparator): The first treatment group received onabotulinumtoxinA (Botox) on the right side of their face and abobotulinumtoxinA (Dysport) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  Interventions: Drug: onabotulinumtoxinA; Drug: abobotulinumtoxinA
- Treatment Arm B (Active Comparator): The second treatment group received abobotulinumtoxinA (Dysport) on the right side of their face and onabotulinumtoxinA (Botox) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  Interventions: Drug: onabotulinumtoxinA; Drug: abobotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — OnabotulinumtoxinA (Botox; Allergan) was approved by the FDA in 2002. Intervention administered by study nurse. Intradermal administered in a regular 1 cm2 grid across the cheeks and forehead. Intramuscular administered as per normal practice.
  Other Names: Botox
Drug: abobotulinumtoxinA — AbobotulinumtoxinA (Dysport; Galderma) was approved by the FDA in 2009. Intervention administered by study nurse. Intradermal administered in a regular 1 cm2 grid across the cheeks and forehead. Intramuscular administered as per normal practice.
  Other Names: Dysport

SUMMARY:
A 16-week single-blind, split-face, randomized study. Each patient served as their own control, receiving onabotulinumtoxinA and abobotulinumtoxinA randomized to either the left or right side of the face. Patients received intradermal BTXA injections at week 0 and intramuscular BTXA injections at week 2. The objective is to examine the effectiveness of intradermal botulinum toxin type A (BTXA) injection in improving skin texture and midface lift while reducing pore size and sebum production, as well as investigate the differences in effectiveness between onabotulinumtoxinA and abobotulinumtoxinA using intradermal and intramuscular injection methods.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between ages of 35 to 65 years (inclusive) who exhibit static wrinkles in the following areas: glabella (forehead frowns), periorbital area (crows feet). Static wrinkles in additional areas of the face are also acceptable.
* Subject is willing to maintain the same skin care regimen throughout the study and has already maintained this skin care regime for 4 weeks prior to baseline.
* The subject is able to comply with study procedures and instructions and is committed to attend all study visits within the given timelines.
* Subject is judged to be a good candidate by study nurse upon identification of dynamic and/or static wrinkles in the areas of movement, and with a moderate amount of skin laxity.
* Subject is willing to use contraception
* A signed informed consent form by a subject able to give consent, prior to any study procedures are performed.

Exclusion Criteria:

* Sensitivity and/or contraindications to botulinum toxin A other ingredients contained in the botulinum toxin A products.
* Any medical condition, in the opinion of the investigator, that would interfere with safety or any study procedures (e.g. auto-immune disease, history of severe allergies, hypertrophic scars, immunotherapeutic treatment, inflammatory or infectious complaints at injection sites, unable to give consent)
* Treatment with botulinum toxin A injections in the neck or face within 1 year of baseline treatment
* Treatment with facial fillers less than 1 year prior to baseline
* Females of childbearing potential who are pregnant, breastfeeding or plan to get pregnant during the course of the study.
* Previous treatment with Lasers, Ultrasound Technology or Radio Frequency on the face and/or neck within 1 year prior to baseline.
* Treatment with Accutane (isotretinoin) or other oral medications for acne during 1 year prior to baseline.
* The use of anti-aging products containing retinol
* Known allergy to cow's milk protein

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Sapra, MD, FRCPC, Principal Investigator — ICLS Dermatology & Plastic Surgery

IPD SHARING:
Plan to Share IPD: Yes
Photographs of individual participants are included in presentations and publications. Consent to reproduce photographs has been obtained from all participants. No other IPD is planned to be shared unless requested.

REFERENCES:
- [Derived] Sapra P, Demay S, Sapra S, Khanna J, Mraud K, Bonadonna J. A Single-blind, Split-face, Randomized, Pilot Study Comparing the Effects of Intradermal and Intramuscular Injection of Two Commercially Available Botulinum Toxin A Formulas to Reduce Signs of Facial Aging. J Clin Aesthet Dermatol. 2017 Feb;10(2):34-44. Epub 2017 Feb 1. PMID 28367260

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm A: The first treatment group received onabotulinumtoxinA (Botox) on the right side of their face and abobotulinumtoxinA (Dysport) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  onabotulinumtoxinA: OnabotulinumtoxinA (Botox; Allergan) was approved by the FDA in 2002. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
  abobotulinumtoxinA: AbobotulinumtoxinA (Dysport; Galderma) was approved by the FDA in 2009. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across
- Treatment Arm B: The second treatment group received abobotulinumtoxinA (Dysport) on the right side of their face and onabotulinumtoxinA (Botox) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  onabotulinumtoxinA: OnabotulinumtoxinA (Botox; Allergan) was approved by the FDA in 2002. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
  abobotulinumtoxinA: AbobotulinumtoxinA (Dysport; Galderma) was approved by the FDA in 2009. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm A: The first treatment group received onabotulinumtoxinA (Botox) on the right side of their face and abobotulinumtoxinA (Dysport) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized. OnabotulinumtoxinA was approved by the FDA in 2002. AbobotulinumtoxinA was approved by the FDA in 2009. Intervention administered by study nurse. Intradermal administered in a regular 1 cm2 grid across the cheeks and forehead. Intramuscular administered according to normal practice.
- Treatment Arm B: The second treatment group received abobotulinumtoxinA (Dysport) on the right side of their face and onabotulinumtoxinA (Botox) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized. OnabotulinumtoxinA was approved by the FDA in 2002. AbobotulinumtoxinA was approved by the FDA in 2009. Intervention administered by study nurse. Intradermal administered in a regular 1 cm2 grid across the cheeks and forehead. Intramuscular administered according to normal practice.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [44 to 60] | 51.1 [51.1 to 60] | 51.1 [51.1 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Blinded assessment of facial rhytids [Mean (Full Range); unit: units on a scale] — 5 point scale. 0=Wrinkles absent (minimum), 1=shallow but visible wrinkles, 2=fine lines slight indentation, 3=clear indentation(0-1mm deep), 4=moderate(1-2mm), 5=deep(>2mm) (maximum). Higher value means a worse outcome (more severe wrinkles). 9 subscales used to obtain 1 score for each patient. Same 5 point scale used for all subscales. Subscales assess different areas of the face. The 9 scales include assessments of the left & right forehead, glabella, around eyes on left & right, left & right cheek, left & right upper lip. Total per patient achieved by taking average of all 9 subscales.
  units on a scale | 2.5 [1.6 to 3] | 2.8 [2.4 to 3] | 2.7 [1.6 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Blinded Assessment: Overall Change in Facial Wrinkles From Baseline to Week 2 as Assessed by a Numeric Rating Scale Based on Pre- and Post-treatment Photographs
Description: Blinded assessments of overall change in facial wrinkles from baseline to week 2 based on pre and post treatment photographs. Measured on a 5 point scale which is a static assessment of wrinkle severity. 0=wrinkles absent (minimum), 1=shallow but visible wrinkles, 2=fine lines slight indentation, 3=clear indentation 0-1mm deep, 4=moderate indentation 1-2mm deep, 5=deep indentation >2mm deep (maximum). A higher value = a worse outcome (more severe wrinkles). Includes 9 subscales measured on the same scale described above. Subscales measure wrinkle severity in the left and right forehead region, left and right cheek region, left and right crow's feet region, left and right upper lip region, and glabellar region. All scores were computed by averaging subscale ratings.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Overall change in wrinkles score. This is calculated per patient, regardless of randomization.
Arm/Group | Arm 1
Number analyzed (Participants) | 10
units on a scale | -0.21 (0.39459)
Statistical Analysis 1: Comparison: Arm 1; Test type: Equivalence — Each variable compared with the "no change" score. The "no change" score is 0 for wrinkles-related variables; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Blinded Assessment: Overall Change in Facial Wrinkles From Baseline to Week 4 as Assessed by a Numeric Rating Scale Based on Pre- and Post-treatment Photographs
Description: Blinded assessments of overall change in facial wrinkles from baseline to week 4 based on pre and post treatment photographs. Measured on a 5 point scale which is a static assessment of wrinkle severity. 0=wrinkles absent (minimum), 1=shallow but visible wrinkles, 2=fine lines slight indentation, 3=clear indentation 0-1mm deep, 4=moderate indentation 1-2mm deep, 5=deep indentation >2mm deep (maximum). A higher value = a worse outcome (more severe wrinkles). Includes 9 subscales measured on the same scale described above. Subscales measure wrinkle severity in the left and right forehead region, left and right cheek region, left and right crow's feet region, left and right upper lip region, and glabellar region. All scores were computed by averaging subscale ratings.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 10
units on a scale | -0.36 (0.419042)
Statistical Analysis 1: Comparison: Arm 1; Test type: Equivalence — Each variable compared with the "no change" score. The "no change" score is 0 for wrinkles-related variables; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Blinded Assessment: Overall Change in Facial Wrinkles From Baseline to Week 16 as Assessed by a Numeric Rating Scale Based on Pre- and Post-treatment Photographs
Description: Blinded assessments of overall change in facial wrinkles from baseline to week 16 based on pre and post treatment photographs. Measured on a 5 point scale which is a static assessment of wrinkle severity. 0=wrinkles absent (minimum), 1=shallow but visible wrinkles, 2=fine lines slight indentation, 3=clear indentation 0-1mm deep, 4=moderate indentation 1-2mm deep, 5=deep indentation >2mm deep (maximum). A higher value = a worse outcome (more severe wrinkles). Includes 9 subscales measured on the same scale described above. Subscales measure wrinkle severity in the left and right forehead region, left and right cheek region, left and right crow's feet region, left and right upper lip region, and glabellar region. All scores were computed by averaging subscale ratings.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 10
units on a scale | -0.3889 (0.440262)
Statistical Analysis 1: Comparison: Arm 1; Test type: Equivalence — Each variable compared with the "no change" score. The "no change" score is 0 for wrinkles-related variables; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 months (September 2013-January 2015)
Groups:
- Treatment Arm A: The first treatment group received onabotulinumtoxinA (Botox) on the right side of their face and abobotulinumtoxinA (Dysport) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  onabotulinumtoxinA: OnabotulinumtoxinA was approved by the FDA in 2002. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
  abobotulinumtoxinA: AbobotulinumtoxinA was approved by the FDA in 2009. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
- Treatment Arm B: The second treatment group received abobotulinumtoxinA (Dysport) on the right side of their face and onabotulinumtoxinA (Botox) on the left side of their face. Baseline treatment at Week 0 included the intradermal injection of onabotulinumtoxinA on one side of the face and abobotulinumtoxinA on the other. Patients were treated at Week 2 with traditional intramuscular injections consisting of onabotulinumtoxinA on the same side of their face as at Week 0 and abobotulinumtoxinA on the other side. Patients were treated based on individual need, and thus the treatment volumes were not controlled or standardized.
  onabotulinumtoxinA: OnabotulinumtoxinA was approved by the FDA in 2002. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
  abobotulinumtoxinA: AbobotulinumtoxinA was approved by the FDA in 2009. Intervention administered by study nurse. Administered in a regular 1 cm2 grid across the cheeks and forehead.
Arm/Group | Treatment Arm A | Treatment Arm B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A (N=5) | Treatment Arm B (N=5)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Mild severity
Drooping (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) — Mild severity
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild severity
Face flushed (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild severity
Pain during injection (Nervous system disorders) | 0 (0) | 1 (1) — Mild severity
Acne breakout (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild severity
Welt on forehead (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Mild severity
Stinging sensation on face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild severity
Itchiness (Nervous system disorders) | 1 (1) | 0 (0) — Mild severity
Left cheek looks more full (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild severity
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) — Mild severity
Worsening inflammation at sacroiliac joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Mild severity
Cold (Immune system disorders) | 0 (0) | 1 (1) — Mild severity
Numbness on forehead (Nervous system disorders) | 0 (0) | 1 (1) — Mild severity

LIMITATIONS AND CAVEATS:
Limitations include small sample size and not having objective assessments. Insignificant p value could mean no difference detected or the sample was too small to detect difference. Blinded assessor made subjective assessments based on the photos.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No